CLINICAL TRIAL: NCT04926532
Title: An Open-label, Single Arm, Multi-center Pilot Study of Programmed Cell Death Protein 1 Antibody (PD-1# Toripalimab Combined With Sorafenib in Patients With Advanced Hepatocellular Carcinoma Cannot Undergo Surgical Resection and TACE
Brief Title: Toripalimab Plus Sorafenib in Patients With Advanced-Stage Hepatocellular Carcinoma
Acronym: Toripalimab
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSGW-PD1-sora
Record Dates: First submitted 2019-10-09; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Toripalimab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — toripalimab; Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab + Sorafenib (Experimental): Toripalimab was administered intravenously at a fixed dose of 240 mg, and the infusion time was 60 ± 5 min, once every 21 days. The cumulative longest medication period is 2 years. Sorafenib was taken orally after meals, twice a day.
  Interventions: Drug: Toripalimab; Drug: Sorafenib

INTERVENTIONS:
Drug: Toripalimab — Toripalimab is a humanized anti-PD-1 monoclonal antibody
Drug: Sorafenib — Sorafenib is a multi-kinase inhibitor

SUMMARY:
Toripalimab is a programmed cell death protein 1 antibody.This is an open-label, single arm, multi-center exploratory study.The objective of this study is to evaluate the efficacy and safety of therapy with toripalimab and sorafenib in patients with advanced stage hepatocellular carcinoma.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy and safety of therapy with toripalimab and sorafenib in patients with advanced stage hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age: 18-75 years old, male or female;
2. Hepatocellular carcinoma diagnosis confirmed by imaging, histopathology or cytology (fibrous layer and mixed hepatocyte/cholangiocarcinoma subtype do not meet the inclusion criteria).
3. According to the clinical stage of Chinese liver cancer (2017 edition), the stage is stage II b or III, and one of the following conditions is met: (1) patients with hepatocellular carcinoma who cannot undergo surgical resection; (2) are unwilling to undergo surgical resection or arterial Patients with hepatocellular carcinoma treated with chemoembolization (TACE).
4. Child-Pugh liver function scores were grade A or B within 7 days prior to the first dose of study drug.
5. Laboratory tests must meet the following criteria within 7 days of starting treatment:

   1. Neutrophils ≥1.5 × 109/L;
   2. platelets ≥ 50 × 109 / L;
   3. hemoglobin ≥ 90g / L (not infused with concentrated red blood cells within 2 weeks);
   4. serum creatinine ≤ 1.5 upper limit of normal (ULN) and creatinine clearance ≥ 50ml / min;
   5. aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN;
   6. serum albumin ≥ 30g / L;
   7. Patients who did not receive anticoagulant therapy: INR ≤ 1.5 × ULN. If the patient receives prophylactic anticoagulant therapy, the INR ≤ 2 × ULN within 14 days before the start of the study treatment and the activated partial thromboplastin time is within the normal range, acceptable for enrollment;
   8. serum bilirubin ≤ 1.25 × ULN;
6. Life expectancy is >3 months.
7. Confirm that there is at least one measurable lesion based on the RECIST 1.1 standard.
8. The Physical Status (PS) score of the Eastern Cooperative Oncology Group (ECOG) was 0-1 within 7 days prior to the first dose of study drug.
9. Male subjects must agree to take contraceptives during treatment and at least 120 days after the last study drug administration, and during this time no sperm can be donated.
10. Female subjects must not be pregnant, not breastfeeding, and at least one of the following conditions can be included in the study: women who do not have fertility or who agree to be at least 120 days after the treatment and the last study drug administration Fertility women who take contraceptive measures as required by the programme.
11. Subject (or legal representative, if applicable) provides informed consent to participate in the study.
12. Subjects with previous or persistent hepatitis C virus (HCV) infection will be eligible to participate in the study. Subjects who are treated must complete treatment at least 1 month before starting the study treatment.
13. Controlled hepatitis B subjects are eligible to participate in the study as long as they meet the following criteria: The HBV viral load must be less than or equal to 10,000 IU/mL prior to the first study drug administration. Subjects receiving anti-HBV therapy with a viral load of less than or equal to 10,000 IU/mL should maintain the same treatment throughout the study treatment period. Anti-hepatitis B core antibody HBc positive, hepatitis B surface antigen (HBsAg) negative, anti-hepatitis B surface antibody (HBsAb) negative or positive, and subjects with HBV viral load below 10000 IU/mL do not need anti- HBV prophylactic treatment.
14. Blood pressure (BP) range of ≤150/90 mm Hg with or without antihypertensive drugs, and the qualification of subjects receiving ≥4 antihypertensive drugs prior to the study will require approval by the sponsor.
15. Subjects have normal organ function, such as thyroid function, pituitary function, and bone marrow function.
16. Specimens must be collected within 7 days prior to initiation of study treatment.

Exclusion Criteria:

1. Esophageal or gastric varices bleeding occurred in the past 6 months.
2. There is a bleeding or thrombotic disease or use an X-factor inhibitor or anticoagulant, such as warfarin or similar, that requires monitoring of the International Normalized Ratio (INR). Treatment with low molecular weight heparin is permitted. Antiplatelet drugs were banned throughout the study.
3. Clinically significant ascites that was not controlled by drugs when examined. (Note: Ascites found only through imaging examinations is allowed to participate in the study)
4. According to imaging examination, there is a tumor thrombus invasion, inferior vena cava or cardiac involvement at the portal vein (Vp4).
5. It has been clinically diagnosed as hepatic encephalopathy in the past 6 months. Subjects with hepatic encephalopathy controlled with rifaximin or lactulose are not allowed to participate in the study.
6. There are medical contraindications that do not accept any contrast-enhanced imaging (CT or MRI).
7. Existing ≥ 3 gastrointestinal or non-gastrointestinal fistulas.
8. Clinically significant hemoptysis or tumor hemorrhage for any cause within 2 weeks prior to the first dose of study drug.
9. Major cardiovascular damage within 12 months prior to the first dose of study drug: a history of congestive heart failure, grade II or older, unstable angina, myocardial infarction, or cerebrovascular accident, or with the New York Heart Association (NYHA) Arrhythmias associated with hemodynamic instability.
10. Suffering from severe unhealed wounds, ulcers or fractures.
11. Previously received any surgery, intervention, radiotherapy, systemic chemotherapy, targeted therapy, anti-PD-1 and anti-PD-L1 antibodies and Chimeric Antigen Receptor T-Cell Immunotherapy and other immunotherapy.
12. Vaccines were administered within 30 days prior to the first dose of study drug. Live vaccines include, but are not limited to, measles, mumps, rubella, varicella/herpes (chickenpox), yellow fever, rabies, Bacillus Calmette Guerin, and typhoid vaccine. Since the seasonal influenza vaccine for injection is usually an inactivated virus vaccine, it is allowed to be used; however, an intranasal influenza vaccine (for example, FluMist) is a live attenuated vaccine and is therefore not allowed.
13. Currently participating in or previously participating in a trial drug study, or using a test device within 4 weeks prior to the first dose of the study drug. Note: Subjects who have entered the clinical trial follow-up period may participate in this trial, provided that the last trial is administered 4 weeks after the last dose of the drug.
14. Diagnosis of immunodeficiency or long-term systemic steroid therapy (daily dose over 10 mg prednisone equivalent) or any form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
15. Another malignant tumor is known and is currently undergoing progress or has been actively treated in the past 3 years. Note: Subjects who have received skin basal cell carcinoma, cutaneous squamous cell carcinoma, or carcinoma in situ (eg, breast cancer, cervical cancer in situ) that may be curable may be treated.
16. A known history or any evidence of central nervous system (CNS) metastasis and/or cancerous meningitis, as assessed by local research center researchers.
17. Those who are severely allergic to research interventions and/or any of their excipients (≥3).
18. Active autoimmune diseases (ie, immunomodulatory drugs, corticosteroids, or immunosuppressive drugs) that require systemic therapy in the past 2 years. Autoimmune diseases such as autoimmune hepatitis, interstitial pneumonia, Uveitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid syndrome-related vascular thrombosis, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, Angiitis, glomerulonephritis, etc., hyperthyroidism or hypothyroidism, asthma requiring bronchodilator treatment, etc., immunomodulatory drugs, corticosteroids or immunosuppressive drugs). Alternative treatments (eg, thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered systemic and are permitted.
19. Clinically significant liver diseases are known, including active viral hepatitis, alcoholic hepatitis or other hepatitis, severe cirrhosis, fatty liver, hereditary liver disease, liver atrophy, portal hypertension, uncontrollable major seizures or Superior vena cava syndrome; for unexplained liver disease, after eliminating viral infection, alcohol and other reasons, it is required to detect autoimmune antibodies and exclude autoimmune liver disease.

    1. Active viral hepatitis is defined as: HBV infection with hepatitis B virus DNA (HBV DNA) > 10000 cps/mL; or HCV infection;
    2. Patients with previous HBV infection or HBV infection who have been cured [defined as hepatitis B virus core antibody (HBcAb) positive and hepatitis B virus surface antigen (HBsAg) negative] may participate in this study. In the first 28 days before administration, the HBV DNA test results of this type of patients must be ≤ 10000 cps/mL;
    3. Patients with positive HCV antibody test results can only be included in the study when the results of polymerase chain reaction (PCR) detection of hepatitis C virus ribonucleic acid (HCV RNA) are negative.
20. The study enrolled with dual active HBV infection (HBsAg (+) and/or detectable HBV DNA) and HCV infection (anti-HCV Ab(+) and detectable HCV RNA.
21. There were dual active HBV infections and hepatitis D virus infections at the time of enrollment.
22. There is a history of (non-infectious) pneumonia requiring steroid therapy or current pneumonia.
23. Urine test strips Subjects with proteinuria >1+ will receive 24-hour urine collection for quantitative assessment of proteinuria. Subjects with urinary protein ≥1 g/24 h were not eligible.
24. Correct QT (QTc) interval extension > 480ms (Fridericia formula correction).
25. Left ventricular ejection fraction (LVEF) measured by multi-gate acquisition scan (MUGA) or echocardiography (ECHO) is below the normal range of the mechanism.
26. Active infections that require systemic therapy, with the exception of HBV and HCV.
27. A history of human immunodeficiency virus (HIV) infection is known. HIV testing is not required unless mandatory by local health authorities.
28. History of active tuberculosis (Bacillus tuberculosis).
29. It is possible to interfere with the test results, the history of the disease or disease evidence, treatment or laboratory values that interfere with the subject's full participation in the study, or the investigator believes that participating in the study is not in the best interest of the subject.
30. Known mental illness or substance abuse conditions can impede the ability of the subject to meet research requirements.
31. During the study period, from the screening visit until 120 days after the last dose of the trial treatment, pregnancy or lactation, or planning to become pregnant or become a father.
32. Subjects who have received allogeneic tissue/solid organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 1 year
  The proportion of patients in this trial whose tumor is destroyed or significantly reduced by the treatment. The extent of the reduction is assessed by researchers based on the RECIST 1.1 standard.

SECONDARY OUTCOMES:
Progression free survival (PFS) | through study completion, an average of 1 year
  The length of time during and after the treatment, that a patient lives with the tumor but it does not get worse.
Disease Control Rate (DCR) | through study completion, an average of 1 year
  The percentage of patients who have achieved complete response, partial response and stable disease after treatment.
Duration of relief (DOR) | through study completion, an average of 1 year
  The length of time that a tumor continues to respond to treatment without the cancer growing or spreading.
Overall survival | 10 year
  Evaluated by patients' survival status

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided